CLINICAL TRIAL: NCT04297033
Title: Lovastatin for Treatment of Brain Arteriovenous Malformations:a Double-blind, Placebo-controlled Randomized Trial
Brief Title: Lovastatin for Treatment of Brain Arteriovenous Malformations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVM-lovastatin
Record Dates: First submitted 2020-02-21; First posted 2020-03-05 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Cerebral Arteriovenous Malformation
Keywords: Cerebral Arteriovenous Malformation, Lovastatin
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lovastatin intervention (Experimental): combination of 40mg/d 12m lovastatin and symptomatic treatment drugs as a treatment strategy for BAVM .
  Interventions: Drug: Lovastatin
- placebo (Placebo Comparator): combination of placebo and symptomatic treatment drugs as a treatment strategy for BAVM
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin — lovastatin 40mg/d 12m
  Arms: Lovastatin intervention
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this pilot study is to evaluate the disease-modifying efficacy of lovastatin in patients with brain arteriovenous malformation.

DETAILED DESCRIPTION:
Brain arteriovenous malformations are lesions that consist of multiple arteries and veins, connecting as a fistula without intervening normal capillary bed. As the disease progresses, the lesion may cause several adverse clinical events including stroke, seizure or even death. For patients with BAVM deemed unsuitable for invasive treatment or who has elected to defer invasive treatment, it is essential to take effective medical management.

Lovastatin possesses antiinflammatory and antiproliferative actions in human endothelial and vascular smooth muscle cells independent of its lipid-lowing action. These findings suggest that lovastatin may be beneficial for maintaining vascular stability, which may contribute to slowing down the progression of the disease and reducing the incidence of adverse clinical events.

The purpose of this pilot study is to evaluate the safety and disease-modifying efficacy of lovastatin in patients with BAVMs. Participants will be randomly assigned to receive either combination of lovastatin and symptomatic treatment drugs or combination of placebo and symptomatic treatment drugs. Patients will have post-dose safety follow-up visit at 1, 3, 6, and 12 months after the study begins. The changes in clinical outcomes, including lesion volume changes and the rate of stroke, seizure or death, will be evaluated in a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have BAVM diagnosed by MRI/MRA, CTA and/or angiogram
2. BAVM deemed unsuitable for invasive treatment OR patient has elected to defer invasive treatment
3. Patient must be 18 years of age or older
4. Sign the informed consent

Exclusion Criteria:

1. Patient has received prior BAVM interventional therapy (endovascular, surgical, radiotherapy)
2. Patient has multiple-foci BAVMs
3. Patient has any form of arteriovenous or spinal fistulas

   Previous diagnosis of any of the following -
4. Patient was diagnosed with Vein of Galen type malformation
5. Patient was diagnosed with cavernous malformation
6. Patient was diagnosed with dural arteriovenous fistula
7. Patient was diagnosed with venous malformation
8. Patient was diagnosed with neurocutaneous syndrome such as cerebro-retinal angiomatosis (von Hippel-Lindau), encephalo-trigeminal syndrome (Sturge-Weber), or Wyburn-Mason syndrome
9. Patient was diagnosed with BAVMs in context of moya-moya-type changes
10. Patient was diagnosed with hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber)
11. Contraindication to an HMG-coA-reductase inhibitor
12. History of adverse reaction to HMG-coA-reductase inhibitors (rhabdomyolysis, hepatitis)
13. Use of any cholesterol lowering medication in the previous 12 weeks

    Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this treatment
14. Impaired liver function with aspartate transaminase (AST) or alanine transaminase (ALT) is more than twice limit of normal.
15. Creatine kinase (CK) is more than twice limit of normal.
16. Medications that interfere with the metabolism of lovastatin
17. Gastrointestinal disease that would affect the ability to swallow or take oral medications or absorb them.
18. End stage renal disease (creatinine clearance eGFR <30 mL/min) or history of severe cardiac disease (angina, myocardial infarction or cardiac surgery in preceding two years)
19. Patient has a history of chronic alcohol or drug abuse within 2 years prior to being recruited
20. Patient has known allergy against iodine contrast agents
21. Patient is pregnant or lactating
22. Inability to provide informed consent.
23. Participation in any clinical investigation within 2 months prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1244 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of stroke between two arms | 24 months
  Stroke is defined as a clinically symptomatic event (any new focal neurological deficit, seizure, or new-onset headache) that is associated with imaging findings of haemorrhage or infarction. Haemorrhage is defined as fresh intracranial blood on head CT or MRI, or in the cerebrospinal fluid. Infarction is defined as a new ischaemic lesion on cranial CT or MRI (diffusion-weighted, T2-weighted, or fluid-attenuated inversion recovery MRI).

SECONDARY OUTCOMES:
Change in AVM volume from baseline MRI | baseline, 6 months, 12 months, 18 months, 24 months
  The volume of arteriovenous malformations will be measured by using MRIcron. The brain arteriovenous malformations will be traced directly on the brain MRIs using MRIcron. Masks of the brain arteriovenous malformations will be drawn on each patient's T1 image in native space by board-certified neurosurgeons, who are blinded to the patients' clinical information. Then, the volume of arteriovenous malformations can be calculated by MRIcron.
Changes in the incidence of seizures and death between two arms | 24 months
  Seizures and death are caused by lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China